CLINICAL TRIAL: NCT02308254
Title: Effects of Lixisenatide on Gastric Emptying, Glycaemia and 'Postprandial' Blood Pressure in Type 2 Diabetes and Healthy Subjects.
Brief Title: Drug Trial of Lixisenatide on Gastric Emptying and Blood Pressure Drops in Type 2 Diabetics and Healthy People
Acronym: Lixi
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Adelaide Hospital (Other)
Collaborators: Sanofi (Industry); National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Karen Jones, Professor, Royal Adelaide Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 130419
Record Dates: First submitted 2014-11-03; First posted 2014-12-04 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus; Gastroparesis
Keywords: Blood pressure; Gastric emptying; Glycemia; Appetite; Incretin Hormones; Superior mesenteric artery blood low
MeSH Terms: conditions — Diabetes Mellitus; Gastroparesis | interventions — lixisenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lixisenatide (Active Comparator): Lixisenatide: 10 mcg, one subcutaneous injection dose
  Interventions: Drug: Lixisenatide
- Placebo (Placebo Comparator): Matching placebo: one subcutaneous injection dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lixisenatide — Abdominal administration
  Other Names: Lyxumia
  Arms: Lixisenatide
Drug: Placebo — Abdominal administration
  Other Names: Dummy
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of the drug lixisenatide on blood sugar levels, stomach emptying, blood pressure and heart rate, release of gut hormones and blood flow in the gut after a glucose drink in both healthy subjects and people with type 2 diabetes. If lixisenatide is shown to be effective, it would encourage ongoing evaluation of its potential use in the management of the falls in blood pressure following a meal in diabetic patients.

DETAILED DESCRIPTION:
Lixisenatide is a drug that has been shown to reduce postprandial glycaemia in people with type 2 diabetes and is now approved for use in Australia. Although slowing of gastric emptying is likely to be the dominant mechanism by which lixisenatide reduces postprandial glycaemia after a meal, the effects of lixisenatide on gastric emptying have hitherto not been quantified by the 'gold standard' technique of scintigraphy. The study would determine and evaluate for the first time the magnitude of, and the relationship between lixisenatide on glycaemia with those on gastric emptying with scintigraphy. This information will be of fundamental significance to the effective use of lixisenatide in the management of people with type 2 diabetes that suffer from postprandial hypotension.

Postprandial hypotension represents an important clinical disorder that occurs frequently in the elderly and people with type 2 diabetes and for which current management is suboptimal. While the mechanisms mediating postprandial hypotension are poorly understood, impaired regulation of splanchnic blood flow, gastric distension, the rate of small intestinal delivery and neural and hormonal mechanisms have been identified as possible pathophysiological mechanisms. Meal ingestion is associated with splanchnic blood pooling and a consequent reduction in venous return of blood to the heart. In healthy young and older individuals, with intact baroreflex mechanisms, these changes induce a rise in heart rate, stoke volume and cardiac output leading to a compensatory rise in blood pressure. However, patients with postprandial hypotension, these responses are inadequate to maintain blood pressure. The magnitude of the fall in blood pressure is greater when gastric emptying is more rapid and that slowing gastric emptying can markedly attenuate the postprandial fall in blood pressure in both healthy older subjects and type 2 patients.

There is currently no information about the effect of lixisenatide on postprandial blood pressure and splanchnic blood flow in patients with type 2 diabetes.

The purpose of this study would determine whether lixisenatide reduces the postprandial fall in blood pressure and related effects of gastric emptying to those on blood pressure, heart rate and splanchnic blood flow.

The use of lixisenatide on appetite and energy intake and how these relate to effects of gastric emptying is lacking.

It is hypothesized that lixisenatide will slow gastric emptying of oral glucose; attenuate both fasting and the postprandial rise in blood glucose; attenuate the magnitude of the fall in blood pressure, rise in heart rate and increase in SMA flow and reduce hunger, increase fullness and decrease energy intake at a buffet meal with greater effects in patients with type 2 diabetes that healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects:

  * Male or female (females using appropriate contraceptive method or willing to undergo pregnancy test)
  * Body Mass Index (BMI) 19 - 30 kg/m2
* Type 2 Diabetic Patients:

  * As per "healthy subjects"
  * Type 2 diabetes (World Health Organisation (WHO) criteria) managed by diet alone or on metformin
  * Glycated haemoglobin >6.0% and <8.5%

Exclusion Criteria:

* Subjects with a history of severe respiratory, cardiovascular, hepatic and/or renal disease (severe in that the social or physical manifestations of the disease, or living with the condition, impact negatively and significantly on the individuals' ability to lead a normal day to day life), chronic alcohol abuse or epilepsy (excluded by history) or if iron status, or liver function tests are outside the following ranges:

  1. Alanine aminotransferase (ALT) 0 - 55 U/L
  2. Alkaline phosphatase 30 - 110 U/L
  3. Aspartate transaminase 0 - 45 U/L
  4. Amylase and/or lipase >3 x ULN
  5. Bilirubin 6 - 24 mmol/L
  6. Ferritin 15 - 200 ng/mL (females); 30 - 300 ng/mL (males)
  7. Haemoglobin 115 - 155 g/L (females); 135 - 172 g/L (males)
* Subjects with a creatinine clearance cut-off of <50 ml/min
* Subjects requiring medication likely to influence blood pressure or gastrointestinal function
* Subjects with a past history of gastrointestinal disease, including known gastroparesis, significant upper gastrointestinal symptoms and previous gastric surgery
* Subjects with a past history of unexplained pancreatitis, chronic pancreatitis, pancreatectomy
* Subjects with a current or prior history of c-cell carcinoma
* Smoking > 10 cigarettes/day
* Alchohol consumption > 20 g/day
* Subjects who have donated blood in the previous 12 weeks
* Women of childbearing potential with no effective contraceptive method (defined as premenopausal, not surgically sterile women for at least 3 months prior to the time of screening) must have a confirmed negative urine B-hCG pregnancy test at screening visit. They must also use an effective contraceptive method throughout the study, and agree to repeat urine pregnancy test at designated visits.
* Lactation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 4.5 hours per study
  Systolic and diastolic blood pressure (mmHg)

SECONDARY OUTCOMES:
Heart rate | 4.5 hours per study
  Heart rate (beats per minute)
Gastric emptying rate | 3 hours per study
  Gastric retention (percent in the total stomach)
Blood glucose concentration | 3 hours per study
  Blood glucose (mmol/L)

OTHER OUTCOMES:
Intragastric distribution | 3 hours per study
  percent retention in the proximal and distal stomach
Gastrointestinal hormone release (concentrations of GLP-1, GIP, C-peptide and 3-OMG) | 4.5 hours per study
  concentrations of GLP-1, GIP, C-peptide and 3-OMG
Superior mesenteric artery blood flow | 3.5 hours per study
  Doppler ultrasound (ml/min)
Appetite (visual analogue questionnaire) | 4.5 hours per study
  sensations of hunger, fullness, desire to eat (mm)
Cardiac output | 3.5 hours per study
  Finapres (L)
Stroke volume | 3.5 hours per study
  Finapres (L)

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Jones, PhD, Principal Investigator — University of Adelaide, Royal Adelaide Hospital
Locations (1):
- Discipline of Medicine, Royal Adelaide Hospital, Adelaide, South Australia, Australia

REFERENCES:
- [Background] Schirra J, Houck P, Wank U, Arnold R, Goke B, Katschinski M. Effects of glucagon-like peptide-1(7-36)amide on antro-pyloro-duodenal motility in the interdigestive state and with duodenal lipid perfusion in humans. Gut. 2000 May;46(5):622-31. doi: 10.1136/gut.46.5.622. PMID 10764704
- [Background] Brennan IM, Feltrin KL, Horowitz M, Smout AJ, Meyer JH, Wishart J, Feinle-Bisset C. Evaluation of interactions between CCK and GLP-1 in their effects on appetite, energy intake, and antropyloroduodenal motility in healthy men. Am J Physiol Regul Integr Comp Physiol. 2005 Jun;288(6):R1477-85. doi: 10.1152/ajpregu.00732.2004. Epub 2005 Feb 3. PMID 15695321
- [Background] Nauck MA, Niedereichholz U, Ettler R, Holst JJ, Orskov C, Ritzel R, Schmiegel WH. Glucagon-like peptide 1 inhibition of gastric emptying outweighs its insulinotropic effects in healthy humans. Am J Physiol. 1997 Nov;273(5):E981-8. doi: 10.1152/ajpendo.1997.273.5.E981. PMID 9374685
- [Background] Little TJ, Pilichiewicz AN, Russo A, Phillips L, Jones KL, Nauck MA, Wishart J, Horowitz M, Feinle-Bisset C. Effects of intravenous glucagon-like peptide-1 on gastric emptying and intragastric distribution in healthy subjects: relationships with postprandial glycemic and insulinemic responses. J Clin Endocrinol Metab. 2006 May;91(5):1916-23. doi: 10.1210/jc.2005-2220. Epub 2006 Feb 21. PMID 16492694
- [Background] Delgado-Aros S, Kim DY, Burton DD, Thomforde GM, Stephens D, Brinkmann BH, Vella A, Camilleri M. Effect of GLP-1 on gastric volume, emptying, maximum volume ingested, and postprandial symptoms in humans. Am J Physiol Gastrointest Liver Physiol. 2002 Mar;282(3):G424-31. doi: 10.1152/ajpgi.2002.282.3.G424. PMID 11841992
- [Background] Horowitz M, Nauck MA. To be or not to be--an incretin or enterogastrone? Gut. 2006 Feb;55(2):148-50. doi: 10.1136/gut.2005.071787. PMID 16407380
- [Background] Horowitz M, Rayner CK, Jones KL. Mechanisms and clinical efficacy of lixisenatide for the management of type 2 diabetes. Adv Ther. 2013 Feb;30(2):81-101. doi: 10.1007/s12325-013-0009-4. Epub 2013 Feb 13. PMID 23423907
- [Background] Riddle M, Home P, Marre M, Niemoeller E, Ping L, Rosenstock J. Efficacy and safety of once-daily lixisenatide in type 2 diabetes insufficiently controlled with basal insulin ± metformin: GetGoal-L Study. Diabetes 2012;61(Suppl 1):A212-A344 (Abstract 983-P).
- [Background] Rosenstock J, Forst T, Aronson R, et al. Efficacy and safety of once-daily lixisenatide added on to titrated glargine plus oral agents in type 2 diabetes: GetGoal-Duo 1 Study. Presented at the 72nd Scientific Sessions of the American Diabetes Association, Philadelphia PA, 8-12 June 2012 (Abstract 62-OR).
- [Background] Ahrén B, Dimas L, Miossec P, Saubado S, Aronson R. Efficacy and safety of lixisenatide QD morning and evening injections vs placebo in T2DM inadequately controlled on metformin (GetGoal-M). Oral presentation at the 21st World Diabetes Congress, Dubai, UAE, 8 December 2011 (Abstract 0-0591).
- [Background] Ratner R, Hanefield M, Shamanna P, et al. Efficacy and safety of lixisenatide once daily versus placebo in patients with T2DM insufficiently controlled on sulfonylurea + metformin (GetGoal-S). Poster presented at 47th Annual Meeting of the European Association for the Study of Diabetes, 12-16 September 2011, Lisbon, Portugal. Diabetologia 2011;54(Suppl 1):1-542 (Abstract 785).
- [Background] Pinget M, Goldenberg R, Niemoeller E, Muehlen-Bartmer I, Guo H, Aronson R. Efficacy and safety of lixisenatide once daily versus placebo in type 2 diabetes insufficiently controlled on pioglitazone (GetGoal-P). Diabetes Obes Metab. 2013 Nov;15(11):1000-7. doi: 10.1111/dom.12121. Epub 2013 May 26. PMID 23627775
- [Background] Rosenstock J, Raccah D, Koranyi L, et al. Efficacy and safety of lixisenatide once daily versus exenatide twice daily in patients with T2DM insufficiently controlled on metformin (GetGoal-X). Poster presented at 47th Annual Meeting of the European Association for the Study of Diabetes, 12-16 September 2011, Lisbon, Portugal. Diabetologia 2011;54(Suppl 1):1-542 (Abstract 786).
- [Background] Bolli G, Munteanu M, Dotsenko S, Niemoeller E, Boka G, Hanefield M. Efficacy and safety of lixisenatide once-daily versus placebo in patients with T2DM insufficiently controlled on metformin (GetGoal-F1). Poster presented at 47th Annual Meeting of the European Association for the Study of Diabetes, 12-16 September 2011, Lisbon, Portugal. Diabetologia 2011;54(Suppl 1): 1-542 (Abstract 784).
- [Background] Fonseca VA, Alvarado-Ruiz R, Raccah D, Boka G, Miossec P, Gerich JE; EFC6018 GetGoal-Mono Study Investigators. Efficacy and safety of the once-daily GLP-1 receptor agonist lixisenatide in monotherapy: a randomized, double-blind, placebo-controlled trial in patients with type 2 diabetes (GetGoal-Mono). Diabetes Care. 2012 Jun;35(6):1225-31. doi: 10.2337/dc11-1935. Epub 2012 Mar 19. PMID 22432104
- [Background] Meier JJ, Kemmeries G, Holst JJ, Nauck MA. Erythromycin antagonizes the deceleration of gastric emptying by glucagon-like peptide 1 and unmasks its insulinotropic effect in healthy subjects. Diabetes. 2005 Jul;54(7):2212-8. doi: 10.2337/diabetes.54.7.2212. PMID 15983224
- [Background] Christensen M, Knop FK, Vilsboll T, Holst JJ. Lixisenatide for type 2 diabetes mellitus. Expert Opin Investig Drugs. 2011 Apr;20(4):549-57. doi: 10.1517/13543784.2011.562191. Epub 2011 Mar 11. PMID 21391833
- [Background] Jansen RW, Lipsitz LA. Postprandial hypotension: epidemiology, pathophysiology, and clinical management. Ann Intern Med. 1995 Feb 15;122(4):286-95. doi: 10.7326/0003-4819-122-4-199502150-00009. PMID 7825766
- [Background] Shannon JR, Diedrich A, Biaggioni I, Tank J, Robertson RM, Robertson D, Jordan J. Water drinking as a treatment for orthostatic syndromes. Am J Med. 2002 Apr 1;112(5):355-60. doi: 10.1016/s0002-9343(02)01025-2. PMID 11904109
- [Background] Vanis L, Gentilcore D, Lange K, Gilja OH, Rigda RS, Trahair LG, Feinle-Bisset C, Rayner CK, Horowitz M, Jones KL. Effects of variations in intragastric volume on blood pressure and splanchnic blood flow during intraduodenal glucose infusion in healthy older subjects. Am J Physiol Regul Integr Comp Physiol. 2012 Feb 15;302(4):R391-9. doi: 10.1152/ajpregu.00464.2011. Epub 2011 Nov 30. PMID 22129616
- [Background] Jones KL, Tonkin A, Horowitz M, Wishart JM, Carney BI, Guha S, Green L. Rate of gastric emptying is a determinant of postprandial hypotension in non-insulin-dependent diabetes mellitus. Clin Sci (Lond). 1998 Jan;94(1):65-70. doi: 10.1042/cs0940065. PMID 9505868
- [Background] O'Donovan D, Feinle C, Tonkin A, Horowitz M, Jones KL. Postprandial hypotension in response to duodenal glucose delivery in healthy older subjects. J Physiol. 2002 Apr 15;540(Pt 2):673-9. doi: 10.1113/jphysiol.2001.013442. PMID 11956353
- [Background] Mathias CJ. Postprandial hypotension. Pathophysiological mechanisms and clinical implications in different disorders. Hypertension. 1991 Nov;18(5):694-704. doi: 10.1161/01.hyp.18.5.694. No abstract available. PMID 1937669
- [Background] Edwards CM, Todd JF, Ghatei MA, Bloom SR. Subcutaneous glucagon-like peptide-1 (7-36) amide is insulinotropic and can cause hypoglycaemia in fasted healthy subjects. Clin Sci (Lond). 1998 Dec;95(6):719-24. doi: 10.1042/cs0950719. PMID 9831697
- [Background] Barragan JM, Rodriguez RE, Eng J, Blazquez E. Interactions of exendin-(9-39) with the effects of glucagon-like peptide-1-(7-36) amide and of exendin-4 on arterial blood pressure and heart rate in rats. Regul Pept. 1996 Nov 14;67(1):63-8. doi: 10.1016/s0167-0115(96)00113-9. PMID 8952007
- [Background] White J. Efficacy and safety of incretin based therapies: clinical trial data. J Am Pharm Assoc (2003). 2009 Sep-Oct;49 Suppl 1:S30-40. doi: 10.1331/JAPhA.2009.09079. PMID 19801363
- [Background] Gentilcore D, Bryant B, Wishart JM, Morris HA, Horowitz M, Jones KL. Acarbose attenuates the hypotensive response to sucrose and slows gastric emptying in the elderly. Am J Med. 2005 Nov;118(11):1289. doi: 10.1016/j.amjmed.2005.05.019. No abstract available. PMID 16271921
- [Background] Stevens JE, Horowitz M, Deacon CF, Nauck M, Rayner CK, Jones KL. The effects of sitagliptin on gastric emptying in healthy humans - a randomised, controlled study. Aliment Pharmacol Ther. 2012 Aug;36(4):379-90. doi: 10.1111/j.1365-2036.2012.05198.x. Epub 2012 Jun 28. PMID 22738299
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Jones KL, MacIntosh C, Su YC, Wells F, Chapman IM, Tonkin A, Horowitz M. Guar gum reduces postprandial hypotension in older people. J Am Geriatr Soc. 2001 Feb;49(2):162-7. doi: 10.1046/j.1532-5415.2001.49037.x. PMID 11207870
- [Background] Gentilcore D, Nair NS, Vanis L, Rayner CK, Meyer JH, Hausken T, Horowitz M, Jones KL. Comparative effects of oral and intraduodenal glucose on blood pressure, heart rate, and splanchnic blood flow in healthy older subjects. Am J Physiol Regul Integr Comp Physiol. 2009 Sep;297(3):R716-22. doi: 10.1152/ajpregu.00215.2009. Epub 2009 Jun 24. PMID 19553500
- [Background] Gentilcore D, Hausken T, Meyer JH, Chapman IM, Horowitz M, Jones KL. Effects of intraduodenal glucose, fat, and protein on blood pressure, heart rate, and splanchnic blood flow in healthy older subjects. Am J Clin Nutr. 2008 Jan;87(1):156-61. doi: 10.1093/ajcn/87.1.156. PMID 18175750
- [Background] Langewouters GJ, Settels JJ, Roelandt R, Wesseling KH. Why use Finapres or Portapres rather than intra-arterial or intermittent non-invasive techniques of blood pressure measurement? J Med Eng Technol. 1998 Jan-Feb;22(1):37-43. doi: 10.3109/03091909809009997. PMID 9491357
- [Background] Moneta GL, Taylor DC, Helton WS, Mulholland MW, Strandness DE Jr. Duplex ultrasound measurement of postprandial intestinal blood flow: effect of meal composition. Gastroenterology. 1988 Nov;95(5):1294-301. doi: 10.1016/0016-5085(88)90364-2. PMID 3049214
- [Background] Iwao T, Toyonaga A, Shigemori H, Oho K, Sumino M, Sato M, Tanikawa K. Echo-Doppler measurements of portal vein and superior mesenteric artery blood flow in humans: inter- and intra-observer short-term reproducibility. J Gastroenterol Hepatol. 1996 Jan;11(1):40-6. doi: 10.1111/j.1440-1746.1996.tb00008.x. PMID 8672740
- [Background] Zwolak RM, Fillinger MF, Walsh DB, LaBombard FE, Musson A, Darling CE, Cronenwett JL. Mesenteric and celiac duplex scanning: a validation study. J Vasc Surg. 1998 Jun;27(6):1078-87; discussion 1088. doi: 10.1016/s0741-5214(98)60010-0. PMID 9652470
- [Background] Shimamoto H, Kito H, Kawazoe K, Fujita T, Shimamoto Y. [Validation of Doppler arterial flow in humans]. Kokyu To Junkan. 1992 Jul;40(7):673-6. Japanese. PMID 1518974
- [Derived] Marathe CS, Pham H, Wu T, Trahair LG, Rigda RS, Buttfield MDM, Hatzinikolas S, Lange K, Rayner CK, Mari A, Horowitz M, Jones KL. Acute Administration of the GLP-1 Receptor Agonist Lixisenatide Diminishes Postprandial Insulin Secretion in Healthy Subjects But Not in Type 2 Diabetes, Associated with Slowing of Gastric Emptying. Diabetes Ther. 2022 Jun;13(6):1245-1249. doi: 10.1007/s13300-022-01258-4. Epub 2022 Apr 22. PMID 35460043